CLINICAL TRIAL: NCT03714841
Title: A Multi-center Randomized Controlled Trial of C-reactive Protein Measurement on Ordering of Blood Cultures in Emergency Department Patients With Sepsis
Brief Title: C-reactive Protein Information and Blood Cultures for Emergency Department Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Rob Stenstrom, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H15-03281
Record Dates: First submitted 2018-03-13; First posted 2018-10-22 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Infection; Bacteremia
Keywords: C reactive protein; randomized controlled trial; Blood culture
MeSH Terms: conditions — Sepsis; Infections; Bacteremia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRP value (Experimental): The patients point of care CRP value is known by the treating physician
  Interventions: Other: CRP
- CRP value unknown (Active Comparator): The patients point of care CRP value is not known by the treating physician
  Interventions: Other: CRP

INTERVENTIONS:
Other: CRP — Knowledge of CRP value

SUMMARY:
Patients with sepsis (2 or more systemic inflammatory response syndrome criteria and suspected infection) assessed in the emergency department have blood cultures obtained to identify potential blood stream infections (BSI). Blood cultures are expensive, sometimes inaccurate, and only positive about 10% of the time in the emergency department.

This study evaluates the effect of physician knowledge of C-reactive protein (CRP) levels on ordering rates of blood cultures in emergency department patients with sepsis. All patients with sepsis will have CRP levels measured using a point-of-care device, prior to blood tests being ordered. Half of participants will have their CRP level available to the emergency physician and half will not. Blood culture ordering rate and safety outcomes will be compared between these two groups.

DETAILED DESCRIPTION:
Sepsis, which is defined as the presence of a systemic inflammatory response syndrome (SIRS) in conjunction with a suspected or proven infection, is a significant cause of morbidity and mortality. It is an extremely common presentation in emergency departments. Most sepsis protocols and guidelines call for blood cultures to be obtained in patients with sepsis, in order to identify blood stream infections (BSI) which are usually caused by bacteria in the blood.

Blood cultures obtained in the emergency department are costly, subject to false positive results, and only positive about 10% of the time. Also, they rarely change patient management.

C-reactive protein (CRP) is an inflammatory marker that rises rapidly in the presence of bacterial infections. Because CRP rises as much as 100 times normal levels in the presence of bacterial infections, we have used it successfully to identify patients with sepsis who do not require a blood blood culture, we believe that physicians knowledge of CRP levels can help to guide their decision to order blood cultures.Patients with sepsis (2 or more SIRS criteria and presumed infection) will have their CRP levels measured using a point of care device (Alere Afinion AS100 Analyzer) prior to blood tests being ordered. Patients will be randomized to either have their CRP value shown to the attending physician or not. Rates of blood culture ordering and safety outcomes will then be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patients with sepsis: Known or presumed infection and 2 or more SIRS criteria: heart rate > 90/minute; respiratory rate > 20/minute; Oral temperature ≥ 38◦ C or < 36◦ C; white blood cell count > 12,000 or < 4,000.
* Able to read and understand consent form in English
* Age 19 years or greater

Exclusion Criteria:

* Patients presenting with septic shock (systolic blood pressure < 90 mmHG)
* Patients at risk for endocarditis (previous episodes of endocarditis, injection drug use)
* Imuno-compromised patients: HIV positive and not on anti-retrovirals; active chemotherapy ; known immune disorder; on immune system modulating drugs, including corticosteroids.
* indwelling venous catheter (dialysis line, Hickman catheter)
* hospitalization in previous 2 weeks
* Surgical procedure in previous 2 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2017-01-21 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Blood culture obtained | 8 hours
  Blood cultures ordered (Yes/No)

SECONDARY OUTCOMES:
28 day mortality | 28 days
  Patient died within 28 days
false positive blood culture | 28 days
  false positive blood culture (Y/N)
Antibiotic prescribing | 7 days
  number of antibiotic prescriptions provided
length of stay | 28 days
  Length of emergency department stay (days)
Admission to hospital | 7 days
  patient admitted to hospital (yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stenstrom, MD, PhD, Principal Investigator — Providence Health & Services
Locations (2):
- Canada (2):
  - St Paul's Hospital, Vancouver, British Columbia
  - Mount St Joseph's Hospital, Vancouver, British Columbia

REFERENCES:
- [Derived] Kyriazopoulou E, Poulakou G, Giamarellos-Bourboulis EJ. Biomarkers in sepsis: can they help improve patient outcome? Curr Opin Infect Dis. 2021 Apr 1;34(2):126-134. doi: 10.1097/QCO.0000000000000707. PMID 33534419